CLINICAL TRIAL: NCT06339580
Title: A Proof-on-concept Study to Investigate the Potential Use of Volume-targeted Ventilation in Patients With Slowly Progressive Neuromuscular Disease
Brief Title: Assessment of Volume-targeted Ventilation in Patients With Neuromuscular Disease
Acronym: VT-NMD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 324456
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VT-NMD arm (Experimental): all patients will be trialed on volume targeted non invasive ventilation
  Interventions: Device: Volume-targeted non-invasive ventilation

INTERVENTIONS:
Device: Volume-targeted non-invasive ventilation — A target tidal volume is set on the ventilation device, and the device will then automatically adjust delivered pressures to reach this target tidal volume.

SUMMARY:
Assessment of safety and efficacy of volume-targeted ventilation in patients with neuromuscular disease.

DETAILED DESCRIPTION:
Patients with neuromuscular diseases (NMD) can suffer from breathing difficulties requiring treatment with a breathing device known as non-invasive ventilation (NIV). NIV aims to support the lungs in removing the waste gas, carbon dioxide (CO2). This is important because patients with high CO2 levels tend to have worse clinical outcomes.

NIV delivers different pressures to the airway when the patient breathes in and when they breathe out. Usually, the pressures it delivers are fixed; i.e. they do not change breath-to-breath. Newer technology allows the machine to independently change the pressures, depending on various patient factors it can measure. There are a small number of studies that suggested that these 'auto-titrating' machines may improve control of carbon dioxide but further work is needed. One of these modes allows us to set a target volume that should be delivered to the patient each breath, and the machine changes settings to deliver this target volume, in response to changing patient parameters. We aim to investigate the safety and efficacy of this volume-targeted NIV (VT-NIV), in order to generate data to design a randomised controlled trial to compare VT-NIV with fixed-NIV.

Patients with NMD who use fixed-NIV will be admitted for a two-night stay to our centre. On the first night, their CO2 control will be assessed on their current ventilator. On the second night, they will be switched to the VT-NIV mode. They will be discharged and asked to use the new mode for three months. Individuals with well-controlled CO2 with their usual mode will allow us to assess the safety of VT-NIV, and individuals with poorly-controlled CO2 will allow us to assess its efficacy. At three months, they will attend an outpatient visit, where use of the new mode will be assessed through data download from the machine and completion of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Slowly progressive neuromuscular disease
* Established on fixed bi-level ventilation
* Documented clinical respiratory stability by supervising clinician (no hospitalizations, respiratory infections or change to ventilator settings in preceding 6 weeks)

Exclusion Criteria:

* Rapidly progressive neuromuscular disease
* Decompensated respiratory failure (pH < 7.35)
* Pregnancy
* Aged <18, >80
* Poor adherence to NIV (<4hrs per night)
* Significant physical or psychiatric co-morbidity that would prevent compliance with trial protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean overnight transcutaneous carbon dioxide | 2 night
  Average carbon dioxide level overnight

SECONDARY OUTCOMES:
Maximum overnight transcutaneous carbon dioxide | 2 night
  Maximum carbon dioxide level reached overnight
Overnight desaturation index | 2 night
  The number of desaturation episodes per night during sleep
Visual analogue scale of sleep comfort | 2 night
  Assessment of sleep comfort on each ventilator on 100mm scale. Min score 0mm (worse sleep comfort), Maximum score 100mm (best sleep comfort)
Health-related quality of life | 3 months
  - Quality of Life Measure for people with slowly progressive and genetic neuromuscular disease questionnaire. Minimum score (worst QoL) 0, Maximum score (best QoL) 100.
Adherence to ventilation | 3 months
  average hours per night the patient uses the ventilator,

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust, London
  - Guy's & St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No